CLINICAL TRIAL: NCT05502783
Title: A Phase II Study Using Fostamatinib to Treat Post-Hematopoietic Stem Cell Transplant Immune-Mediated Cytopenias
Brief Title: Using Fostamatinib to Treat Post-Hematopoietic Stem Cell Transplant Immune-mediated Cytopenias
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Clinical trial was halted prematurely due to low enrollment
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000758; 000758-H
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Immune Mediated Anemia; Immune Mediated Thrombocytopenia; Chronic GVHD
Keywords: Allogeneic Hematopoietic Stem Cell Transplant; Graft Versus Host Disease; Spleen Tyrosine Kinase (Syk) Inhibitor
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Bronchiolitis Obliterans Syndrome; Graft vs Host Disease | interventions — fostamatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fostamatinib in Participants Post-Hematopoietic Stem Cell Transplant with Immune-Mediated Cytopenias (Experimental): Participants Post-Hematopoietic Stem Cell Transplant with Immune-Mediated Cytopenias will receive fostamatinib 100 mg BID by mouth for 4 weeks. On the 4-week evaluation, a) if cytopenia improves (hemoglobin =10 g/dL, platelets = 50 x 109/L), patients will continue the same dose for a total of 12 weeks, b) if refractory cytopenias persist (hemoglobin < 10 g/dL, platelets < 50 x 109/L), the dose will be increased to 150 mg BID. Subjects with persistent (=2 readings, 2 weeks apart) loss of hematologic response after week 5 can increase their dose to 150 mg BID until at end of the study on week 12.
  Interventions: Drug: fostamatinib

INTERVENTIONS:
Drug: fostamatinib — Participants will receive fostamatinib 100 mg BID for 4 weeks. On the 4-week evaluation, a) if cytopenia improves (hemoglobin =10 g/dL, platelets = 50 x 109/L), patients will continue the same dose for a total of 12 weeks, b) if refractory cytopenias persist (hemoglobin < 10 g/dL, platelets < 50 x 109/L), the dose will be increased to 150 mg BID. Subjects with persistent (=2 readings, 2 weeks apart) loss of hematologic response after week 5 can increase their dose to 150 mg BID until at end of the study on week 12.

SUMMARY:
Background:

People who have a blood stem cell transplant can sometimes develop cytopenia. This means that their levels of one or more types of blood cell, such as the red cells or platelets, are lower than they should be. This can occur because a person s immune system might attack these cells after a stem cell transplant. Cytopenia can lead to anemia, severe bleeding, infections, and other problems. Treatments are needed to help keep blood cell levels stable after blood stem cell transplant.

Objective:

To test a study drug (fostamatinib) in people who have cytopenia after a blood stem cell transplant.

Eligibility:

People aged 18 to 75 years who have cytopenia after a blood stem cell transplant.

Design:

Participants will be screened. They will have a physical exam. They will have blood, urine, and stool tests.

Fostamatinib is an oral tablet taken by mouth. Participants will take the pills 2 times a day for 12 weeks.

Participants will have a medical assessment every 2 weeks; their vital signs will be checked, and they will have blood and stool tests. Participants must come to the NIH clinic for these visits in weeks 4 and 12. Other visits may be done by telephone or telehealth; the blood and stool tests can be sent to the researchers from a local lab.

After 4 weeks, some participants may begin taking a higher dose of the drug.

Participants will return for a final medical assessment 2 weeks after they finish taking the drug.

Participants who complete this study and show evidence that fostamatinib has increased their blood cell counts may enroll in an extension study to continue taking fostamatinib.

DETAILED DESCRIPTION:
Study Description:

This open label phase II trial is designed to evaluate the efficacy of fostamatinib in the treatment of post-transplant cytopenias as assessed by hematologic improvement in anemia and/or thrombocytopenia following a 12-week treatment course. Patients who respond to the 12-week treatment course on this single arm study are eligible and have the option to enroll on the extended access trial.

Objectives:

The primary objective is to assess efficacy of fostamatinib for stable hematologic recovery during post-hematopoietic stem cell transplant immune mediated anemia and/or thrombocytopenia.

The secondary objective is to assess efficacy of fostamatinib for clinically-relevant outcomes in post-hematopoietic stem cell transplant patients.

The exploratory objective is to evaluate changes in serologic markers that may be associated with cytopenias while on treatment to identify key elements for fostamatinib response.

Endpoints:

Primary endpoints:

The proportion of subjects with hematologic recovery that is stable, defined as improvement documented in 2 consecutive available readings at least 2 weeks apart, without recent blood product transfusion support in the past 7 days.

-Hematologic recovery is defined as:

--Hemoglobin >=10 g/dL (or at least >=2 g/dL above baseline) in subjects enrolled with posttransplant anemia. In subjects with symptomatic anemia, a hemoglobin increase of at least >=2 g/dL above baseline is required

OR

--Platelets >= 50 x 10^9/L (or at least >=20 x 10^9/L above baseline) in subjects enrolled with posttransplant thrombocytopenia

OR

--Both of the above criteria in subjects with posttransplant Evans syndrome

Secondary endpoints:

-Proportion of subjects who achieve objective hematologic recovery within the 12-week treatment course defined as:

--Hemoglobin >=9 g/dL (or at least >=1 g/dL above baseline) in subjects enrolled with anemia or at least >=1 g/dL above baseline in subjects with symptomatic anemia

OR

--Platelets >= 30 x 10^9/L (or at least >=10 x 10^9/L above baseline) in subjects enrolled with thrombocytopenia

OR

-- Either of the above criteria in subjects with Evans syndrome

* Average weekly requirement of transfused blood component or growth factor requirement (total units of PRBC or Platelets/week, total dose of growth factor/week) by week 12, compared to the week prior to the start of the study drug.
* Change in corticosteroid dose over time, measured by median daily weight-based prednisone-equivalent corticosteroid dose in a week, from week 1 to week 12
* Change in other immunosuppressant dose over time, measured by median daily dose of the immunosuppressant in a week, from week 1 to week 12
* Number of patients who achieved >=50% steroid dose reduction by week 12 compared to week 1
* Incidence and severity of cGVHD according to 2014 NIH Consensus Criteria, at baseline before the initiation of treatment, and at week 12

Exploratory endpoints:

* Absolute percentage change in B cell chimerism pre-treatment, vs weeks 4 and 12.
* cPRA change in the preformed HLA antibodies before and after treatment in subjects with thrombocytopenia or Evans syndrome
* Percent MFI change of preformed HLA antibodies before and after treatment. This applies for antibodies with an MFI >1,000.
* Anti-RBC alloantibody titer change in patients with hemolytic anemia before and after treatment
* Assessment of serial cytokines pre-treatment and weeks 4 and 12. Cytokines include CRP, IL-1, IL-2, IL-6, IFN gamma, TNF alpha, EPO and TPO
* Immunoglobulin level changes pre-treatment, and weeks 4 and 12.
* Absolute reticulocyte count, lactate dehydrogenase, haptoglobin changes pre-treatment, and at each biweekly study visit, in patients with anemia or Evans syndrome
* Change in the weekly rate and severity of bleeding according to the total score of the ITP-Bleeding Scale (IBLS), from week -1 (one week before the start of the study drug) to week 12, in subjects with thrombocytopenia or Evans syndrome

ELIGIBILITY:
* INCLUSION CRITERIA:
* Ages 18-75 years inclusive
* Ability to comprehend the investigational nature of the study and provide informed consent
* Female patients of reproductive potential agree to avoid pregnancy through abstinence or the use two forms of highly effective birth control during and for 1 month after the last study treatment and agree not to donate eggs during this time
* male patients of reproductive potential agree to avoid pregnancy of a partner through abstinence or the use two forms of highly effective birth control during and for 1 month after the last study treatment and agree not to donate sperm during this time.
* Diagnosis of an immune mediated cytopenia (anemia and/or thrombocytopenia) in a patient that either:

  * Failed or relapsed after at least one line of therapy including steroids, IVIG, TPO mimetics, rituximab, azathioprine, cyclophosphamide, cyclosporine, tacrolimus, danazol, vincristine, ESA or splenectomy
  * Or remains transfusion dependent (>=1 transfusion(s)/2 weeks)
  * Or is steroid dependent
* Subjects are >=60 days post-allogeneic transplant with:

  * Thrombocytopenia, defined as average platelets count <30 x 10^9/L for 3 consecutive available readings at least 2 weeks apart, after other cell lines have engrafted, with no counts >40 x 10^9/L unless from rescue transfusions. Subjects failed at least one line of therapy outlined above with a clinical diagnosis of immune mediated thrombocytopenia.
  * Anemia, transfusion dependent, or defined as hemoglobin <=9 g/dL for 3 consecutive available readings at least 2 weeks apart, after other cell lines have engrafted OR if hemoglobin 9-10 g/dL, subject must have symptomatic anemia or ongoing treatment for immune hemolytic anemia that have failed at least one line of therapy outlined above. Symptomatic anemia is defined as anemia with fatigue, weakness, shortness of breath, palpitations/fast heartbeat, lightheadedness, and/or chest pain, and these symptoms are attributed to anemia. Laboratory evaluation are recommended but not required for the diagnosis, such as a positive DAT, low haptoglobin <lower limit of normal (LLN), indirect bilirubin > upper limit of normal (ULN), or lactate dehydrogenase (LDH) >ULN.
* Subjects must test negative for HIV, HBV, and HCV by standard serologic tests within the previous six months
* Subjects on other standard of care therapeutic regimens for GVHD or cytopenias should be on a stable dose of medication (no change >=25%) for at least 15 days prior to enrollment.
* Patients with a history of hypertension should be maintained on a stable antihypertensive regimen and with controlled blood pressure (Systolic blood pressure < 140 mmHg and diastolic blood pressure <90 mmHg) for at least one week prior to enrollment.
* Peripheral blood or bone marrow T-cell chimerism >=50% donor cells
* Immune mediated anemia in subjects with auto or alloantibodies identified due to ABO or non-ABO mismatch transplant, or thrombocytopenia due to identified HLA/HPA antibody. Other causes of immune mediated cytopenias include clinically diagnosed (with or without serologic confirmation) idiopathic thrombocytopenic purpura or autoimmune hemolytic anemia. Subjects with cytopenias attributable to GVHD will be included. Subjects with idiopathic immune mediated cytopenias can also be included. Subjects with evidence for graft rejection per the investigator's opinion ARE NOT eligible for treatment.

Steroid dependence is defined as inability to tolerate a corticosteroid taper after demonstrating a response to an initial corticosteroid dose (typically 1-2 mg/kg/day). Patients will meet our definition of steroid dependence if their cytopenias relapse or progress before achieving a 50% decrease in the initial corticosteroid dose and/or are unable to have their steroid dose tapered to a dose of less than 20 mg/day of prednisone.

EXCLUSION CRITERIA:

* Severe psychiatric illness or mental deficiency sufficient to make making informed consent impossible
* Positive pregnancy test for women of childbearing age within 1 week or being actively lactating
* Immune mediated cytopenia responsive to the standard of care treatment
* Immune mediated cytopenia due to other autoimmune causes, such as systemic lupus erythrocytosis, chronic lymphocytic leukemia
* Patients who have previously received or currently take fostamatinib post-allogeneic transplant
* Non-immune mediated cytopenias. Etiologies including, but not limited to, cytopenias due to HIV infection, lymphoproliferative disorders, myelodysplasia/acute leukemia, drug-induced thrombocytopenia, thrombotic microangiopathies, acute bleeding, consumptive coagulopathy, fever, infections leading to cytopenia, medications induced cytopenias, thrombotic microangiopathies (disseminated intravascular coagulation), splenomegaly or hemophagocytic lymphohistiophagocytosis, relapse of primary disease.
* Patients with neutropenia, defined as absolute neutrophil count <=1.0 x 10^9/L, will be excluded
* Uncontrolled hypertension (systolic blood pressure >=140mmHg or diastolic blood pressure >=90mmHg)
* ALT or AST >=3 times the upper limit of normal, or direct bilirubin >=2 times the upper limit of normal
* Patients who have a history of medical disorders, that in the investigator's opinion, could affect the conduct of the study or the absorption, metabolism or excretion of the study drug are excluded.
* Patients with lymphoma/chronic lymphocytic leukemia, hepatitis, or HIV associated with ITP/wAIHA
* Patients with evidence of graft rejection (based on clinical suspicion supported by BM biopsy data and/or chimerism studies and/or MLR)
* Subjects recently treated (within 30 days) with cytokine-targeting biologics (anti-TNF, IL6) or Bcell or plasma-cell depleting antibody.
* Other cancers except that for which the transplant was done < 2 years before study entry, except non-melanoma skin cancer or carcinoma in situ of the uterine cervix or breast

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Y Hur, D.O., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000758-H.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fostamatinib in Participants Post-Hematopoietic Stem Cell Transplant With Immune-Mediated Cytopenias
Started | 1
Completed | 0
Not Completed | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fostamatinib in Participants Post-Hematopoietic Stem Cell Transplant With Immune-Mediated Cytopenias
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Able to Maintain Hematologic Recovery
Description: Stable hematologic recovery (improvement documented in 2 consecutive available readings) without recent blood product transfusion support (in the past 48-72 hours).
  Hematologic recovery is defined as:
  * Hemoglobin =10 g/dL (or at least =2 g/dL above baseline) in participants enrolled with posttransplant anemia. In participants with symptomatic anemia, a hemoglobin increase of at least =2 g/dL above baseline is required OR
  * Platelets = 50 x 10^9/L (or at least =20 x 10^9/L above baseline) in participants enrolled with posttransplant thrombocytopenia OR
  * Both of the above criteria in participants with posttransplant Evans syndrome
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10
Population: One participant withdrew at week 10 from the study due to lack of efficacy, therefore no data was collected up to week 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib in Participants Post-Hematopoietic Stem Cell Transplant With Immune-Mediated Cytopenias
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Number of Participants Who Achieve Objective Hematologic Recovery
Description: Objective hematologic recovery defined as:
  * Hemoglobin =9 g/dL (or at least =1 g/dL above baseline) in participants enrolled with anemia or at least =1 g/dL above baseline in participants with symptomatic anemia OR
  * Platelets = 30 x 10^9/L (or at least =20 x 10^9/L above baseline) in participants enrolled with thrombocytopenia OR
  * Both of the above criteria in participants with Evans syndrome
Time Frame: Up to 10 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib in Participants Post-Hematopoietic Stem Cell Transplant With Immune-Mediated Cytopenias
Number analyzed (Participants) | 1
Participants | 0

3. Secondary Outcome: Median Change in Requirement of Transfused Blood Component
Description: Median change in requirement of weekly transfused blood component or growth factor injections requirement (total units of Packed Red Blood Cells or Platelets). Data from the specified time points were aggregated and summarized to calculate the median value.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Units
Arm/Group | Fostamatinib in Participants Post-Hematopoietic Stem Cell Transplant With Immune-Mediated Cytopenias
Number analyzed (Participants) | 1
Units
  Packed Red Blood Cells | 1.0 [1.0 to 1.0]
  Platelet | 12.0 [12.0 to 12.0]

4. Secondary Outcome: Median Change in Requirement of Growth Factor Injections
Description: Median change in requirement of weekly growth factor injections. Data from the specified time points were aggregated and summarized to calculate the median value.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10
Population: as for outcome 1
Measure: Median (Full Range); unit: Number of Growth Factor Injections
Arm/Group | Fostamatinib in Participants Post-Hematopoietic Stem Cell Transplant With Immune-Mediated Cytopenias
Number analyzed (Participants) | 1
Number of Growth Factor Injections | 1.0 [0 to 1]

5. Secondary Outcome: Median Change in Requirement Corticosteroid Dose (Prednisone)
Description: Median Change in requirement corticosteroid dose (Prednisone) , measured by median daily weight-based prednisone-equivalent corticosteroid dose from week 1 to week 12. Data from the specified time points were aggregated and summarized to calculate the median value.
Time Frame: Baseline, Week 2, Week 4, Week , Week 8, Week 10
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Fostamatinib in Participants Post-Hematopoietic Stem Cell Transplant With Immune-Mediated Cytopenias
Number analyzed (Participants) | 1
mg | 5 [5 to 5]

6. Secondary Outcome: Median Change in Other Immunosuppressant Dose
Description: Median Change in other immunosuppressant dose, measured by median daily dose of the immunosuppressant. Data from the specified time points were aggregated and summarized to calculate the median value.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Population: Participant was not on immunosuppressants during this study, therefore data could not be collected
Arm/Group | Fostamatinib in Participants Post-Hematopoietic Stem Cell Transplant With Immune-Mediated Cytopenias
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants Who Developed Mild, Moderate or Severe Chronic Graft vs Host Disease (GVHD) According to 2014 NIH Consensus Criteria
Description: Number of Participants Who Developed Mild, Moderate or Severe Chronic Graft vs Host Disease (GVHD) according to 2014 NIH Consensus Criteria
  Diagnosis is based on organ involvement and severity scoring, with criteria for skin, mouth, eyes, liver, lungs, gastrointestinal tract, joints/fascia, and genital tract, though criteria have been revised to exclude findings clearly attributable to non-GVHD causes. Severity is categorized as mild, moderate, or severe based on the number of organs involved and the specific severity score for each organ (0-3), with lungs requiring specific pulmonary function tests for scoring.
  Mild: Involves 1 or 2 organs with a score of no more than 1 for each (lung score must be 0).
  Moderate: Involves 3 or more organs with a score of no more than 1 for each; OR at least 1 organ (not the lung) has a score of 2; OR the lung score is 1.
  Severe: Involves at least 1 organ with a score of 3; OR the lung score is 2 or 3.
Time Frame: Up to 10 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib in Participants Post-Hematopoietic Stem Cell Transplant With Immune-Mediated Cytopenias
Number analyzed (Participants) | 1
Participants
  Mild | 0
  Moderate | 0
  Severe | 0

8. Secondary Outcome: Number of Patients Who Achieved 50% Steroid Dose Reduction
Description: Number of patients who achieved 50% steroid dose reduction by week 12 compared to week 1
Time Frame: Up to Week 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib in Participants Post-Hematopoietic Stem Cell Transplant With Immune-Mediated Cytopenias
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: up to 10 weeks
Arm/Group | Fostamatinib in Participants Post-Hematopoietic Stem Cell Transplant With Immune-Mediated Cytopenias
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fostamatinib in Participants Post-Hematopoietic Stem Cell Transplant With Immune-Mediated Cytopenias (N=1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (4)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Generalied edema (General disorders) | 1 (1)
Haptoglobin decreased (Investigations) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (4)
Hyponatremia (Metabolism and nutrition disorders) | 1 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (6)
Pain (General disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/83/NCT05502783/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT05502783/ICF_001.pdf